CLINICAL TRIAL: NCT04035499
Title: A Mobile Health Exercise Intervention for Older Patients With Myeloid Neoplasms
Acronym: GO-EXCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS19090
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Intervention

STUDY DESIGN:
Intervention Model Description: Evaluating the feasibility of a mobile health exercise intervention in older adults with myeloid neoplasms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm:single (Experimental): GO-EXCAP Mobile App involves the use of a mobile app delivery platform to deliver an exercise program [Exercise for Cancer Patients (EXCAP©®)]. EXCAP©® is a progressive walking and resistance exercise program
  Interventions: Behavioral: GO-EXCAP Mobile App

INTERVENTIONS:
Behavioral: GO-EXCAP Mobile App — A mobile app delivery platform and the EXCAP©® exercise program

SUMMARY:
This is a pilot study to evaluate the feasibility of a mobile health exercise intervention (GO-EXCAP Mobile App) over 7 weeks in 25 patients with myeloid neoplasms receiving hypomethylating agents.

DETAILED DESCRIPTION:
Up to 98% of older patients with myeloid neoplasms experience physical function decline, fatigue, and mood disturbances. Mobile health exercise interventions are promising strategy to prevent physical function decline and improve fatigue and mood disturbances, but older patients with myeloid neoplasms receiving hypomethylating agents are understudied. The proposed study will evaluate a novel mobile health exercise intervention that is adapted to older patients with myeloid neoplasms receiving outpatient hypomethylating agents and investigate whether and how exercise can prevent physical function decline, improve fatigue and mood disturbances, and prevent worsening quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age is greater than or equal to 60 years
* Have a diagnosis of MN
* Receiving outpatient chemotherapy (e.g., HMA)
* English speaking
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* No medical contraindications for exercise per oncologist
* Able to walk 4 meters as part of Short Physical Performance Battery measured walk (with or without assistive device)
* Able to provide informed consent

Exclusion Criteria

Platelet count of 10,000 per microliter or less in the most recent blood draw (due to risk of spontaneous bleeding) prior to transfusion (i.e., patients are allowed to enroll if their platelet count is 10,000 per microliter or less but is scheduled to receive transfusion the day of consent)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will also make this protocol available to NIH and NCI at the time of submission of each progress report and at the end of the final funding year. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing.Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion.

REFERENCES:
- [Result] Loh KP, Kleckner IR, Lin PJ, Mohile SG, Canin BE, Flannery MA, Fung C, Dunne RF, Bautista J, Culakova E, Kleckner AS, Peppone LJ, Janelsins M, McHugh C, Conlin A, Cho JK, Kasbari S, Esparaz BT, Kuebler JP, Mustian KM. Effects of a Home-based Exercise Program on Anxiety and Mood Disturbances in Older Adults with Cancer Receiving Chemotherapy. J Am Geriatr Soc. 2019 May;67(5):1005-1011. doi: 10.1111/jgs.15951. PMID 31034591
- [Result] Loh KP, Ramsdale E, Culakova E, Mendler JH, Liesveld JL, O'Dwyer KM, McHugh C, Gilles M, Lloyd T, Goodman M, Klepin HD, Mustian KM, Schnall R, Mohile SG. Novel mHealth App to Deliver Geriatric Assessment-Driven Interventions for Older Adults With Cancer: Pilot Feasibility and Usability Study. JMIR Cancer. 2018 Oct 29;4(2):e10296. doi: 10.2196/10296. PMID 30373733
- [Derived] Jensen-Battaglia M, Lin PJ, Sanapala C, Watson EE, Mendler JH, Liesveld J, Wang Y, Hayward E, LoCastro M, Mortaz S, Dunne RF, Mustian K, Loh KP. Changes in muscle performance among older adults with myeloid malignancies engaging in a mobile health (mHealth) exercise intervention: a single arm pilot study. BMC Geriatr. 2025 Jan 9;25(1):22. doi: 10.1186/s12877-024-05668-w. PMID 39789445
- [Derived] Wang K, Consagra W, Jensen-Battaglia M, Kleckner A, Kleckner IR, Loh KP. Chemotherapy-related symptoms and exercise adherence in older patients with myeloid neoplasms. Support Care Cancer. 2023 Sep 12;31(10):572. doi: 10.1007/s00520-023-08039-0. PMID 37698745
- [Derived] Loh KP, Sanapala C, Watson EE, Jensen-Battaglia M, Janelsins MC, Klepin HD, Schnall R, Culakova E, Vertino P, Susiarjo M, Lin PJ, Mendler JH, Liesveld JL, Huselton EJ, Taberner K, Mohile SG, Mustian K. A single-arm pilot study of a mobile health exercise intervention (GO-EXCAP) in older patients with myeloid neoplasms. Blood Adv. 2022 Jul 12;6(13):3850-3860. doi: 10.1182/bloodadvances.2022007056. PMID 35320340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm:Single
Started | 25
Completed | 22
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Older adults aged 60 and over
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Short Physical Performance Battery at Baseline [Mean (Standard Deviation); unit: score on a scale] — Changes in physical function measured using the Short Physical Performance Battery (SPPB) which an objective physical assessment evaluating lower extremity physical function (score ranges from 0-12; higher score indicates better physical function). It is comprised of 3 components: a four-meter walk, repeated chair stands and a balance test (the score for each component ranges from 0-4). Population: Post-intervention data were not collected for 3 subjects who completed baseline (2 died, 1 withdrew)
  score on a scale
    number analyzed (Participants) | 22
    (all) | 9.0 (1.7)
Brief Fatigue Inventory at Baseline [Mean (Standard Deviation); unit: score on a scale] — Changes in fatigue measures using the Brief Fatigue Inventory (BFI) which is a 9-item, patient-reported instrument. The score for each item ranges from 0-10, a higher score indicates higher self-reported levels of fatigue. Population: Post-intervention data were not collected for 3 subjects who completed baseline (2 died, 1 withdrew)
  score on a scale
    number analyzed (Participants) | 22
    (all) | 29.4 (20.8)
Center for Epidemiologic Studies Depression at Baseline [Mean (Standard Deviation); unit: score on a scale] — Changes in depression measured using the Center for Epidemiological Studies Depression Scale (CES-D) which is a 20-item depression scale. The score for each item ranges from 0-3, a higher score indicates higher self-reported depression levels. Population: Post-intervention data were not collected for 3 subjects who completed baseline
  score on a scale
    number analyzed (Participants) | 22
    (all) | 11.7 (7.7)
Functional Assessment of Cancer Therapy-Leukemia at Baseline [Mean (Standard Deviation); unit: score on a scale] — Changes in quality of life measured using the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) scale. It consists of 44 items divided into 5 subscales: physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), functional well-being (FWB) and leukemia-specific concerns. The score for each item ranges from 0-4. After reversing the scoring of negatively worded items, all the scores are summated. A higher score indicates better quality of life. Population: Measure Analysis Population Description: Post-intervention data were not collected for 3 subjects who completed baseline (2 died, 1 withdrew)
  score on a scale
    number analyzed (Participants) | 22
    (all) | 123.9 (24.7)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Percentage of Patients Entering Any Exercise Data Into the Mobile App ≥50% of the Study Period Days, Excluding Hospitalization
Description: Percentage of patients entering any exercise data into the mobile app ≥50% of the study period days, excluding hospitalization
Time Frame: 8-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
Participants
  % Entering Step Data | 18
  % Entering Resistance Data | 14

2. Primary Outcome: Feasibility: Percentage of Patients Entering Resistance Data Into the Mobile App ≥50% of the Study Period Days, Excluding Hospitalization
Description: Percentage of Patients Entering Resistance Data Into the Mobile App ≥50% of the Study Period Days, Excluding Hospitalization
Time Frame: 8-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
Participants | 14

3. Primary Outcome: Feasibility: Recruitment Rates
Description: Recruitment rates (percentage of patients who are approached and subsequently consent).
Time Frame: Week 0, prior to baseline
Population: Number of potential subjects determined eligible and approached to consent. Patients who consented and subsequently withdrew before baseline assessments also contributed to the numerator.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 59
Participants | 38

4. Primary Outcome: Feasibility: Retention Rates
Description: Retention rates (percentage of patients who are enrolled i.e., complete baseline assessments and subsequently complete post-intervention assessments)
Time Frame: 8-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 25
Participants | 22

5. Secondary Outcome: Pre-post Changes in Short Physical Performance Battery (SPPB)
Description: Changes in physical function measured using the Short Physical Performance Battery (SPPB) which an objective physical assessment evaluating lower extremity physical function (total score ranges from 0-12; higher score indicates better physical function). It is comprised of 3 components: a four-meter walk, repeated chair stands and a balance test (the score for each component ranges from 0-4; scores are summed).
Time Frame: Baseline, Post-Intervention, Changes from baseline to post-intervention (an average of 8-12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
score on a scale
  Baseline | 9.0 (1.7)
  Post-Intervention | 9.2 (2.4)
  Changes from baseline to post | 0.2 (1.6)

6. Secondary Outcome: Pre-post Changes in Brief Fatigue Inventory (BFI)
Description: Changes in fatigue measures using the Brief Fatigue Inventory (BFI) which is a 9-item, patient-reported instrument. The score for each item ranges from 0-10 (scores are summed; total score ranges from 0-90), a higher score indicates higher self-reported levels of fatigue.
Time Frame: Baseline, Post-Intervention, Changes from baseline to post-intervention (an average of 8-12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
score on a scale
  Baseline | 29.4 (20.8)
  Post-Intervention | 23.2 (18.8)
  Changes from baseline to post | -6.2 (17.9)

7. Secondary Outcome: Pre-post Changes in the Center for Epidemiological Studies Depression Scale (CES-D)
Description: Changes in depression measured using the Center for Epidemiological Studies Depression Scale (CES-D) which is a 20-item depression scale. The score for each item ranges from 0-3 (scores are summed; total score ranges from 0-60), a higher score indicates higher self-reported depression levels.
Time Frame: 8-12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
score on a scale
  Baseline | 11.7 (7.7)
  Post-Intervention | 11.1 (8.0)
  Changes from Baseline to Post | -0.6 (6.1)

8. Secondary Outcome: Pre-post Changes in Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu)
Description: Changes in quality of life measured using the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) scale. It consists of 44 items divided into 5 subscales: physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), functional well-being (FWB) and leukemia-specific concerns. The score for each item ranges from 0-4 (total score ranges from 0-176). After reversing the scoring of negatively worded items, all the scores are summated. A higher score indicates better quality of life.
Time Frame: Baseline, Post-Intervention, Changes from baseline to post-intervention (an average of 8-12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Arm:Single
Number analyzed (Participants) | 22
score on a scale
  Baseline | 123.9 (24.7)
  Post-Intervention | 127.1 (22.9)
  Changes from baseline to post | 3.2 (18.1)

ADVERSE EVENTS:
Time Frame: 8-12 weeks
Arm/Group | Experimental Arm:Single
All-Cause Mortality (participants affected / at risk) | 2/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT04035499/Prot_SAP_000.pdf